CLINICAL TRIAL: NCT00119496
Title: A Clinical Study to Investigate the Effect of Rosiglitazone, Theophylline and Inhaled Corticosteroid, Inflammation and Pulmonary Function in Asthmatic Smokers
Brief Title: Rosiglitazone Versus Theophylline in Asthmatic Smokers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: GlaxoSmithKline (Industry); Chest, Heart and Stroke Association Scotland (Other); Chief Scientist Office of the Scottish Government (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES104033; 2004-004247-22 EUDRACT
Record Dates: First submitted 2005-07-01; First posted 2005-07-13 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2007-11

CONDITIONS: Asthma
Keywords: Corticosteroid; Rosiglitazone; Theophylline; Beclomethasone; Inflammation; Asthma; Smoking; Pulmonary
MeSH Terms: conditions — Asthma; Inflammation; Smoking | interventions — Rosiglitazone; Theophylline; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): Inhaled beclomethasone (400mcg/day)
  Interventions: Drug: beclomethasone
- Arm 2 (Active Comparator): Rosiglitazone
  Interventions: Drug: rosiglitazone
- Arm3 (Active Comparator): Oral theophylline
  Interventions: Drug: theophylline
- Arm 4 (Active Comparator): Oral theophylline and inhaled beclomethasone
  Interventions: Drug: inhaled beclomethasone and oral theophylline

INTERVENTIONS:
Drug: rosiglitazone — oral tablet, 4mg bd for 4 weeks
  Other Names: Rosiglitazone Maleate, Avandia
  Arms: Arm 2
Drug: theophylline — Oral theophylline, 200mg bd
  Other Names: uniphyllin
  Arms: Arm3
Drug: beclomethasone — inhaled beclomethasone, 200mcg bd
  Other Names: Qvar
  Arms: Group 1
Drug: inhaled beclomethasone and oral theophylline — inhaled beclomethasone (400mcg/day), oral theophylline (400mg/day)
  Other Names: Qvar and uniphyllin
  Arms: Arm 4

SUMMARY:
Asthmatic smokers display a blunted response to both inhaled and oral corticosteroid treatments and are at increased risk for exacerbations and near fatal asthma. The prevalence of smoking in asthmatics runs between 20-30%. Therefore, new, more efficacious treatments are required.

Recent work has demonstrated a mechanism which may explain steroid resistance. A commonly used drug called theophylline can reverse this steroid resistance in laboratory studies. Another commonly used drug, rosiglitazone can reverse smoking induced lung inflammation in laboratory studies.

The investigators aim to study the effects of these drugs on smoking asthmatics' lung function and other parameters including quality of life and asthma control.

DETAILED DESCRIPTION:
Smoking asthmatics have chronic pulmonary inflammation that is relatively steroid resistant. PPAR agonists (of which rosiglitazone is one example) have been shown to reduce several markers of inflammation in humans and in smoking animal models.

This clinical study will use smoking asthmatics as a human model of smoke-induced steroid-insensitive airway inflammation to evaluate both efficacy of rosiglitazone as an anti-inflammatory drug as well as the effect of low doses of theophylline on the response to low-dose inhaled corticosteroid (LD ICS).

Mild or moderate (as per GINA guidelines) persistent-asthmatic smokers will be randomised into this study after a 4-week washout period during which they will be withdrawn from inhaled corticosteroids (ICS). Subjects will then receive one of four treatments for 28 days: rosiglitazone, LD ICS, theophylline, or LD ICS plus theophylline.

The effects of rosiglitazone and LD ICS on pulmonary function will be compared as a primary objective. In addition, effects of theophylline plus LD ICS will be compared against theophylline and LD ICS separately. Both pulmonary anti-inflammatory and systemic anti-inflammatory activity will also be investigated.

Subjects will have baseline assessments of pulmonary function, biomarkers of systemic inflammation, sputum, exhaled breath biomarkers, asthma control questionnaires and safety parameters. Following 28 days of treatment, these parameters will all be reassessed in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 60 years of age (inclusive).
* Clinical diagnosis of mild or moderate persistent asthma in accordance with the Global Initiative for Asthma (GINA) criteria
* Have had a history of asthma for a minimum of 6 months prior to entry into the study
* Subjects must be current cigarette smokers with a minimum five-pack-year smoking history
* Baseline FEV1 that is greater than 50% predicted; and reversibility of 12% or more at screening, washout or randomisation.
* Capable of providing signed written informed consent and complying with all the specified study procedures.

Exclusion Criteria:

* Asthma exacerbation or a respiratory tract infection within four weeks of screening.
* Type 1 or type 2 diabetes mellitus.
* Women who are lactating, pregnant, or planning to become pregnant.
* Clinically significant renal or hepatic laboratory values (e.g. AST/ALT/total bilirubin/AP > 2.5 times normal values).
* Anaemia (< 11 g/dL for males or < 10 g/dL for females)
* Contraindications to treatment as outlined in any of the product labels
* Prior history of severe oedema or serious fluid related event (e.g., heart failure) associated with any TZD
* The subject has a history of significant hypersensitivity to study drugs
* Presence of unstable or severe angina or congestive heart failure (NYHA class III/IV) or evidence or history of known congestive heart failure (NYHA class I-IV) or an abnormal electrocardiogram (ECG), as determined by the Investigator, or subjects who have had new cardiac events (such as MI, new CHF, PTCA, CABG) within 6 months of screening.
* History or suspicion of current drug abuse or alcohol abuse within the last 6 months.
* History suggestive of active infection or non-asthma lung pathology
* Clinically significant renal disease, metabolic syndrome, cirrhosis (Child-Pugh Class B/C), hypertension or any other clinically significant cardiovascular, neurological, endocrine, or haematological abnormalities that are uncontrolled on permitted therapy.
* Risk factors for human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection at Screening (Visit 1)
* Subjects who are morbidly obese, defined as having a body mass index (BMI) > 40 kg/m2
* Unable to perform spirometry
* Subjects who require treatment with any of the following asthma medications from Screening (Visit 1) until study completion:

  * Inhaled cromolyn sodium or nedocromil;
  * Ipratropium bromide;
  * Xanthines (theophylline preparations);
  * Leukotriene modifiers;
  * Long-acting inhaled beta2-agonists (salmeterol, formoterol);
  * Oral beta2-agonists.
* Treatment with oral, intravenous or intra-articular corticosteroids within 6 weeks of Screening or thereafter.
* Subjects who have been taking in excess of 1000 μg daily of beclomethasone (or equivalent) within 6 weeks of Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2005-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Comparison of pre-bronchodilator (FEV1) at 28 days between rosiglitazone and LD ICS treatment groups. | 28 days

SECONDARY OUTCOMES:
Rosiglitazone vs LD ICS on other endpoints of pulmonary function in smoking asthmatics. | 28 days
Theophylline plus LD ICS vs LD ICS on pulmonary function in smoking asthmatics. | 28 days
Theophylline plus LD ICS vs theophylline on pulmonary function in smoking asthmatics. | 28 days
Safety and tolerability of rosiglitazone, LD ICS, theophylline and theophylline plus LD ICS in smoking asthmatics. | 28 days
To assess the effects in smoking asthmatics of rosiglitazone, LD ICS, theophylline and theophylline plus LD ICS on asthma control using the ACQ (Juniper et al, 1999). | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Thomson, MD, Principal Investigator — University of Glasgow
Locations (1):
- Asthma Research Group, Gartnavel General Hospital, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Background] Spears M, McSharry C, Thomson NC. Peroxisome proliferator-activated receptor-gamma agonists as potential anti-inflammatory agents in asthma and chronic obstructive pulmonary disease. Clin Exp Allergy. 2006 Dec;36(12):1494-504. doi: 10.1111/j.1365-2222.2006.02604.x. PMID 17177672
- [Derived] Spears M, Donnelly I, Jolly L, Brannigan M, Ito K, McSharry C, Lafferty J, Chaudhuri R, Braganza G, Adcock IM, Barnes PJ, Wood S, Thomson NC. Effect of low-dose theophylline plus beclometasone on lung function in smokers with asthma: a pilot study. Eur Respir J. 2009 May;33(5):1010-7. doi: 10.1183/09031936.00158208. Epub 2009 Feb 5. PMID 19196814
- See also: Asthma Research Unit website — http://www.gla.ac.uk/departments/immunology/respiratorymedicine/